CLINICAL TRIAL: NCT03513068
Title: Portable Oxygen Concentrator Improvements to Physical Activity, Oxygen Usage, and Quality of Life in Chronic Obstructive Pulmonary Disease Patients Using Long-term Oxygen Therapy (POC-STEP)
Acronym: POC-STEP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: ResMed (Industry)
Collaborators: Inogen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-16-05-02
Record Dates: First submitted 2018-04-11; First posted 2018-05-01 (Actual); Results first posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2021-09

CONDITIONS: COPD
Keywords: COPD; POC; Oxygen; QoL
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard Of Care (SOC) (No Intervention): Standard of care long-term oxygen therapy
- SOC + POC (Portable Oxygen Concentrator) (Experimental): Standard of care long-term oxygen therapy + POC
  Interventions: Device: Portable Oxygen Concentrator (POC)

INTERVENTIONS:
Device: Portable Oxygen Concentrator (POC) — COPD patients prescribed with LTOT will be randomized to receive a portable oxygen concentrator (POC)
  Arms: SOC + POC (Portable Oxygen Concentrator)

SUMMARY:
To evaluate changes in activity based on the use of portable oxygen concentrators combined with standard of care (SOC) long- term oxygen therapy versus SOC long-term oxygen therapy alone at 12 weeks in patients with COPD who require continuous (24/7) long-term oxygen therapy. The study will also assess oxygen usage, quality of life, hospitalizations and death.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 40 years or older.
2. Patient has a documented diagnosis of COPD.
3. Patient qualifies for continuous (24/7) long-term oxygen therapy.
4. Patient is prescribed oxygen at ≤ 5 L/min.
5. Patient is POC-naïve, i.e., has not used a POC prior to enrolling in this study.
6. Patient is able to tolerate pulsed oxygen therapy, i.e., oxygen delivered via a POC.
7. Patient is able to fully understand study information and provide signed informed consent and HIPAA authorization.

Exclusion Criteria:

1. Patient's condition is contraindicated for the use of a POC.
2. Patient has uncontrolled or untreated sleep-disordered breathing that is uncontrolled or untreated.
3. Patient is unable to complete the 6-minute walk test.
4. Patient has a diagnosis (within less than two weeks prior to study entry) of pneumonia or respiratory infection, and/or acute bronchitis requiring antibiotics, or new/increased dose of systemic corticosteroids.
5. Patient has had thoracic surgery or another procedure in the six months prior to enrollment that is likely to cause instability of pulmonary status.
6. Patient has an open skin ulcer or rash where the activity monitor will be worn on the body.
7. Patient has a life expectancy < 1 year.
8. Patient has non-COPD lung disease that may affect oxygenation or survival.
9. Patient has a planned intervention(s) requiring hospitalization within the three months of study participation.
10. Patient is pregnant or planning to become pregnant.
11. Patient is participating in a clinical study of a medical product and has not completed the required follow-up period.
12. Patient, in the opinion of the investigator, should be excluded from the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2020-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MaryKay Sobcinski, Study Chair — RCRI
Locations (11):
- United States (11):
  - National Jewish Health, Denver, Colorado
  - University of Illinois, Chicago, Chicago, Illinois
  - St. Vincent Airways, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Kentucky Research Group, Louisville, Kentucky
  - ClinSite LLC, Ann Arbor, Michigan
  - Minnesota Lung Center, Edina, Minnesota
  - Minnesota Lung Center, Minneapolis, Minnesota
  - Minnesota Lung Center, Woodbury, Minnesota
  - Sierra Clinical Research, Las Vegas, Nevada
  - UPMC Emphysema/COPD Research Center, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Of Care (SOC) | SOC + POC (Portable Oxygen Concentrator)
Started | 54 | 54
Completed | 49 | 48
Not Completed | 5 | 6
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 4 | 6

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were collected from all participants who signed the ICF; some of these participants did not complete the First study visit.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Of Care (SOC) | SOC + POC (Portable Oxygen Concentrator) | Total
Number analyzed (Participants) | 50 | 46 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (7.9) | 70.2 (9.7) | 68.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 25 | 56
  Male | 19 | 21 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 44 | 43 | 87
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 46 | 96
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.7 (7.8) | 30.7 (7.4) | 30.2 (7.6)

OUTCOME MEASURES:

1. Primary Outcome: Physical Activity Level
Description: Change in physical activity level (PAL) as measured through actigraphy. Outcome measure is the change between the value at Week 12 and Day 1 (Baseline). Min = 0; Max = infinite. A large positive change would indicate the participant increased their activity level at 12 weeks in comparison to Day 1. Physical activity level (PAL) is the ratio of total energy expenditure (TEE) to sleep energy expenditure (SEE). TEE is the total number of wear-filtered kilocalories expended in a day and SEE is the total number of sleep- and wear-filtered kilocalories expended in a day.
Time Frame: 12 weeks
Population: Includes only patients that had evaluable PAL data (via ActiGraph watch) at both baseline and 12 weeks.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Standard Of Care (SOC) | SOC + POC (Portable Oxygen Concentrator)
Number analyzed (Participants) | 40 | 31
Ratio | 14.6 (232.1) | -84.6 (1949.7)

2. Secondary Outcome: St. George Respiratory Questionnaire (SGRQ)
Description: Change in total SGRQ score between Week 12 and Baseline (Day1 ). Measures quality of life in patients with airway obstruction. Scores range from 0 to 100, with higher scores indicating more limitations.
Time Frame: 12 weeks
Population: Includes only patients with evaluable and complete SGRQ data at both Baseline and Week 12.
Measure: Mean (Standard Deviation); unit: score on a scale SGRQ
Arm/Group | Standard Of Care (SOC) | SOC + POC (Portable Oxygen Concentrator)
Number analyzed (Participants) | 48 | 45
score on a scale SGRQ | 1.1 (12.4) | -1.3 (9.1)

3. Secondary Outcome: Oxygen Usage
Description: Change in Total Hours of Use
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Standard Of Care (SOC) | SOC + POC (Portable Oxygen Concentrator)
Number analyzed (Participants) | 46 | 43
hours | 0.4 (2.5) | -0.1 (3.1)

4. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS): Anxiety
Description: Outcome measure is the change from Baseline (Day 1) and Week 12. HADS questionnaire measures anxiety and depression. A patient can score between 0-21, scores of less than 7 indicate non-cases.
Time Frame: 12 weeks
Population: Only includes patients with complete HADS data at both Baseline and Week 12.
Measure: Mean (Standard Deviation); unit: score on a scale HADS
Arm/Group | Standard Of Care (SOC) | SOC + POC (Portable Oxygen Concentrator)
Number analyzed (Participants) | 48 | 45
score on a scale HADS | 0.8 (4.1) | -0.5 (3.0)

ADVERSE EVENTS:
Time Frame: Duration of the study = 12 weeks.
Description: All AEs were collected during the course of the study. Events were categorized as hospitalizations or exacerbations of COPD, respiratory-related event, or Other. Trial sites and Investigators were allowed to capture non-categorized events as "Other".
Arm/Group | Standard Of Care (SOC) | SOC + POC (Portable Oxygen Concentrator)
All-Cause Mortality (participants affected / at risk) | 1/54 | 0/54
Serious Adverse Events (participants affected / at risk) | 6/54 | 1/54
Other Adverse Events (participants affected / at risk) | 21/54 | 16/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Of Care (SOC) (N=54) | SOC + POC (Portable Oxygen Concentrator) (N=54)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (3)
Other respiratory-related condition (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Other (General disorders) | 1 (1) | 1 (7)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Of Care (SOC) (N=54) | SOC + POC (Portable Oxygen Concentrator) (N=54)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 14 (15) | 10 (12)
Other respiratory-related condition (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (3)
Other (General disorders) | 7 (9) | 9 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/68/NCT03513068/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-18): https://cdn.clinicaltrials.gov/large-docs/68/NCT03513068/SAP_001.pdf